CLINICAL TRIAL: NCT03673618
Title: Soluble Corn Fiber Supplementation for Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Collaborators: Northern Arizona University (Other); Flinn Foundation (Unknown); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Phoenixchildrens-18-121
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2022-04

CONDITIONS: Asthma in Children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A study pharmacist will provide soluble corn fiber or a placebo (malodextrin) in identical packets to be dispensed in identical fruit-flavored beverage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROMOTIR soluble corn fiber (Experimental): Participants will ingest PROMOTIR soluble corn fiber (85% fiber, 12 g/day) in a fruit-flavored beverage for 4 weeks alongside their normal diet and normal asthma treatments.
  Interventions: Drug: Soluble Corn Fiber
- Malodextrin (Placebo Comparator): Participants will ingest malodextrin in a fruit-flavored beverage for 4 weeks alongside their normal diet and normal asthma treatments.
  Interventions: Drug: Soluble Corn Fiber

INTERVENTIONS:
Drug: Soluble Corn Fiber — Fiber or placebo

SUMMARY:
Studies of the importance of the human microbiome have demonstrated that microbial metabolites of fermentation of our dietary products (e.g. dietary fiber) have a multitude of health benefits. The investigators aim to determine whether supplementation of asthmatic children with soluble corn fiber alongside standard of care reduces airway inflammation driven by the gut microbial metabolites acetate, propionate, or butyrate (short chain fatty acids).

DETAILED DESCRIPTION:
Asthma is a complex inflammatory disease of the airways that is estimated to affect 300 million people worldwide. Incidence of asthma is steadily increasing in Western populations; an additional 100 million asthma diagnoses are anticipated by the year 2025. Asthma is a multifactorial disease affected by genetic and environmental factors. One major and potentially modifiable environmental factor is the Western diet. The Western diet influences the microbiome, which in turn, may influence inflammatory airway diseases via a gut microbiome-airway connection. The investigators hypothesize that prebiotic dietary fiber supplementation leads to increased circulating short chain fatty acid production and improvement in asthma disease activity. The investigators will recruit 20 children, ages 6-17 years old, with asthma from the Severe Asthma Clinic or General Pulmonary Clinic at Phoenix Children's Hospital. Participants will be randomly assigned (1:1) using a random number generator to ingest PROMOTIR soluble corn fiber (85% fiber, 12 g/day) in a fruit-flavored beverage or placebo (malodextrin in a similar fruit-flavored beverage) as previously described. Participants will be asked to consume the prebiotic soluble corn fiber (or placebo) for 4 weeks alongside their normal diet and normal asthma treatments. Blood will be collected pre- and post-fiber intervention to measure baseline and post-intervention circulating SCFAs. Stool samples and nasal wash will be collected for microbiome and immune analysis pre- and post- fiber consumption. Nasal washes will be collected pre- and post-fiber consumption to measure inflammatory patterns.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma
* Fractional excretion of exhaled nitric oxide (FeNO) > 50 ppb OR a history of environmental allergies
* No emergency department or hospital visits for asthma in the past 3 months
* No systemic corticosteroids in the past 1 month
* Ability to consume a liquid drink of SCF or placebo
* Ability to return for a 4-6 week follow-up visit
* No special or unique diet as determined by PI/CO-Is.

Exclusion Criteria:

* Cystic fibrosis
* Bronchiectasis
* Change in asthma medicines other than short acting bronchodilators planned over the next 4-6 weeks.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Asthma symptoms | 4 weeks
  Asthma Control Questionnaire

SECONDARY OUTCOMES:
Change in Serum Short Chain Fatty Acids | Before treatment period and after treatment for 4 weeks
Change in nasal wash Th2 gene expression | Before treatment period and after treatment for 4 weeks
Alpha and beta diversity in participants' nasal microbiome | Before treatment period and after treatment for 4 weeks
Alpha and beta diversity in participants' stool microbiome | Before treatment period and after treatment for 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix Childrens Hospital, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Rank MA, Barroso DL, Conn KA, Pecak M, Scandura M, Hirsch AH, Gu H, Whisner CM, Shearer H, Johnson D, Argel N, Bauer CS, Williams SN, Wright BL, Woodward J, Cope EK. A randomized, double-blind, placebo-controlled trial of soluble corn fiber supplementation for children with asthma. Front Allergy. 2026 Jan 21;6:1707834. doi: 10.3389/falgy.2025.1707834. eCollection 2025. PMID 41647190